CLINICAL TRIAL: NCT00196040
Title: Feasibility Study of the PFX Closure System in Subjects With Cryptogenic Stroke, Transient Ischemic Attack, Migraine or Decompression Illness
Brief Title: The Paradigm II Trial: PFX Closure System in Subjects With Cryptogenic Stroke, Transient Ischemic Attack, Migraine or Decompression Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cierra (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Foramen Ovale, Patent
MeSH Terms: conditions — Foramen Ovale, Patent

INTERVENTIONS:
Device: PFX Closure System

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of the PFX Closure System when utilized for patent foramen ovale (PFO) in patients suffering from cryptogenic stroke (undetermined cause of stroke), transient ischemic attack (brief neurological dysfunction), migraine or decompression illness.

DETAILED DESCRIPTION:
Patent Foramen Ovale has been implicated in the etiology of paradoxical embolism, cryptogenic stroke, transient ischemic attack, and right to left gas embolism in severe decompression illness. An association between patent foramen ovale and severe migraine headaches has also been reported. Several implantable devices are being used for percutaneous closure of patent foramen ovale; we propose to use a non-implantable system to safely effect closure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 65 years old
* Documented patent foramen ovale as determined by positive micro bubble study demonstrating right to left shunt and/or anatomic detection and functional assessment by pre-operative transcranial Doppler (TCD) and peri-operative echocardiography or ultrasound.
* Subjects with one or more of the following:

  * history of cryptogenic stroke, transient ischemic attack (TIA) or embolism due to presumed paradoxical embolism through a PFO; or
  * history of severe migraine headaches, despite attempted treatment with available migraine medications, for whom other specific causes of migraine headache, such as underlying disease or medications, have been ruled out; or
  * history of severe decompression illness.
* Negative pregnancy test in women who are of child-bearing potential
* Signed Informed Consent form

Additional Inclusion Criteria for Migraine Subjects:

* Onset of migraine before age of 50 years
* History of migraine > 1 year
* Migraine frequency greater than 1 migraine per month

Exclusion Criteria:

* Presence of thrombus at the intended site of closure, in left atrial appendage, or documented evidence of venous thrombus in the vessels through which access to the PFO is gained.
* Active endocarditis, or other infections producing a bacteremia
* Presence of atrial septal defect(s) or fenestrations which allow shunting
* Presence of implanted cardiac valves, pacemakers, cardioverters/defibrillators (ICDs) or vena cava filters.
* Subjects with coagulation disorders or bleeding disorders including gastric ulcers, who are unable to take antiplatelet or anticoagulant therapy
* Subjects with an intra-cardiac mass, tumor, clots or vegetation
* Large, redundant atrial septal aneurysm that would prohibit adequate device access to the PFO or closure of the PFO, in the judgment of the investigator. A coexisting redundant atrial septal aneurysm is considered large if it prohibits the ability of the operator to adequately achieve vacuum suction necessary to achieve PFO closure.
* Presence of conduction abnormality requiring pharmacologic or electrical therapy intervention or 1st degree block
* Current enrollment in any investigational trial(s) using devices implanted in the vascular system or enrolled in any experimental drug study(ies) within three months of study entry
* Religious or other beliefs which would prevent subjects from following all physician directed instructions or prevent compliance with protocol required medications and follow-ups.
* Hemodynamic instability or shock
* History of diabetes requiring treatment with insulin

Additional Exclusion Criteria for Cryptogenic Stroke Subjects:

* History of stroke or TIA within the past 14 days
* Source of stroke other than paradoxical embolization

Additional Exclusion Criteria for Migraine Subjects:

* Seizure disorder
* Other organic central nervous system disease
* Headache as a result of traumatic head or neck injury
* Evidence of alcohol, drug or substance abuse within the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
PFO closure as measured by transesophageal echocardiography (TEE) or intracardiac echocardiography (ICE) acutely post procedure

SECONDARY OUTCOMES:
PFO closure as measured by TEE or transthoracic echocardiography (TTE) at 30 days, 3 or 6 months and 12 months post procedure
Adverse event (AE) rates for all subjects
New conduction abnormality rate through final follow-up
Measurement of migraine severity or frequency at 6 and 12 months post procedure for subjects enrolled due to diagnosis of migraine

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — Cardio Vasculares Centrum - Sankt Katharinen
Locations (1):
- Cardiovascular Center Frankfurt Sankt katharinen, Frankfurt, Germany